CLINICAL TRIAL: NCT05678621
Title: A Randomised Controlled Trial of Continuing Immunoglobulin Therapy, or Stopping With or Without Prophylactic Antibiotics, on Infection Rate in Patients With Acquired Hypogammaglobulinemia Secondary to Haematological Malignancies.
Brief Title: Role of Antibiotic Therapy or Immunoglobulin On iNfections in hAematoLogy: Immunoglobulin Stopping or Extension
Acronym: RATIONALISE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Erica Wood, Professor Erica Wood, Head, Transfusion Research Unit, Public Health and Preventive Medicine, Monash University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRU-RLS-21
Record Dates: First submitted 2022-02-11; First posted 2023-01-10 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Haematological Malignancy; Hypogammaglobulinemia
Keywords: Myeloma; Lymphoma; Leukaemia; Blood cancer; Malignancy; Infection; Antibiotic; Anti-infective agent; Immunoglobulin
MeSH Terms: conditions — Hematologic Neoplasms; Agammaglobulinemia; Neoplasms, Plasma Cell; Lymphoma; Leukemia; Neoplasms; Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Amoxicillin; Clavulanic Acid; Ciprofloxacin; Immunoglobulins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Infectious outcomes and adverse events will be adjudicated by an independent, blinded outcome adjudication committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ARM A: Stop immunoglobulin (Ig) and commence prophylactic oral antibiotics (Experimental): Once daily trimethoprim-sulfamethoxazole (co-trimoxazole) 160mg/800mg. Nb: Doxycycline 100mg daily as an alternative for participants with hypersensitivity to co-trimoxazole.
  Duration: 12 months. Route: PO
  Interventions: Drug: trimethoprim-sulfamethoxazole (co-trimoxazole)
- ARM B: Stop immunoglobulin (without prophylactic antibiotics) (Experimental): Participants will be prescribed amoxycillin/clavulanic acid 1750-2000mg/250mg and ciprofloxacin 750 mg, to keep at home for initial use if symptoms of infection develop, with immediate review by their treating clinical team, or nearest emergency department or medical practitioner with phone contact to treating team if most practical.
  Nb: clindamycin 600 mg is permitted as an alternative to amoxycillin/clavulanic acid for participants with hypersensitivity to penicillin.
  Duration: 12 months. Route: PO
  Interventions: Drug: amoxycillin/clavulanic acid and ciprofloxacin
- ARM C: Continue immunoglobulin (Active Comparator): Participants will continue treatment with their current Ig replacement schedule. Participants will receive either Intravenous Ig (IVIg) or Subcutaneous Ig (SCIg)
  * IVIg: Participants will be treated in accordance with the Criteria for Clinical Use of Immunoglobulin in Australia. Monthly (every 4 weeks ± 1 week) dose of 0.4g/kg, modified to achieve an Immunoglobulin G (IgG) trough level of at least lower limit of age-specific serum IgG reference range. In the first month of therapy, if IgG <4g/L then an additional (loading) dose of 0.4g/kg may be given at the clinician's discretion.
  * SCIg: Subcutaneous immunoglobulin weekly may be used in patients who meet local criteria for home based self-administration in centres with established SCIg programs. A loading IVIg dose may be given in the first month if required. Thereafter, dosing at 100mg/kg/week, modified to achieve an IgG steady state level of at least the lower limit of the serum reference range.
  Duration: 12 months.
  Interventions: Drug: Immunoglobulins

INTERVENTIONS:
Drug: trimethoprim-sulfamethoxazole (co-trimoxazole) — Doxycycline is an alternative for participants with hypersensitivity to co-trimoxazole.
  Arms: ARM A: Stop immunoglobulin (Ig) and commence prophylactic oral antibiotics
Drug: amoxycillin/clavulanic acid and ciprofloxacin — clindamycin is an alternative to amoxycillin/clavulanic acid for participants with hypersensitivity to penicillin.
  Arms: ARM B: Stop immunoglobulin (without prophylactic antibiotics)
Drug: Immunoglobulins — Intravenous monthly immunoglobulin or subcutaneous weekly immunoglobulin
  Arms: ARM C: Continue immunoglobulin

SUMMARY:
The aim of the study is to find out if patients with blood cancers receiving immunoglobulin (Ig) for the purpose of preventing infections can safety stop immunoglobulin after six months of therapy, and take oral antibiotics instead to prevent serious infections.

Patients may be eligible to join this study if they are aged 18 years or above, have an acquired hypogammaglobulinaemia secondary to a haematological malignancy, and have been receiving intravenous or subcutaneous Ig for longer than 6 consecutive months.

Participants will be randomised (allocated by chance) to one of three treatment groups, as follows:

* Stop immunoglobulin (IVIg or SCIg) and be given oral antibiotics to take every day (ARM A)
* Stop immunoglobulin (IVIg or SCIg) and be given oral antibiotics to keep at home to use as soon as symptoms of an infection develop (ARM B)
* Continue receiving immunoglobulin (IVIg or SCIg) - this is the usual care group (ARM C)

The duration of each treatment is for 12 months from study entry.

Participants will be asked to attend a screening/baseline visit so that their treating clinician can assess their eligibility for the trial and collect baseline data. If eligible for the trial, participants will then be randomly allocated to one of the three treatment groups.

Once randomised, active participation in the study will last for 13 months. During this period, participants will be asked to return to the hospital for a study visit every 3 months, with monthly telephone visits to check-in on your progress between each in-person visit. Participants will also be asked to complete a study diary, recording treatment compliance and signs/symptoms of infection experienced throughout the study period.

Types of assessments and data collected will include: Medical history, demographics, physical examination, blood tests, stool sample, quality of life questionnaires, information about your general health, hospitalisations, medications and procedures. In order to assess and compare the cost-effectiveness of the treatment groups, the study team will also request authorisation from participants to access their Medicare Benefits Schedule (MBS), Pharmaceutical Benefits Scheme (PBS), and Australian Immunisation Register (AIR) data.

ELIGIBILITY:
Inclusion Criteria:

1. Aged greater than or equal to 18 years of age
2. Diagnosis of chronic lymphocytic leukaemia (CLL), multiple myeloma (MM) or non-Hodgkin lymphoma (NHL).
3. Patients must be receiving Ig (IV or subcutaneous - SCIg) replacement for prevention of bacterial infections due to hypogammaglobulinaemia for longer than 6 consecutive months.
4. Patient is eligible for trial of Ig cessation in the opinion of the treating clinician and local investigator.
5. Life expectancy greater than 12 months.
6. Able to give informed consent, and willing and able to comply with each of the treatment arms.

Exclusion Criteria:

1. Prior or planned allogeneic haematopoietic stem cell transplantation.
2. Major infection (Grade 3 or higher) in preceding 3 months, and/or current active infection requiring antimicrobial treatment.
3. Already receiving daily antibiotic prophylaxis for the purpose of preventing bacterial infection (Note: patients may receive antiviral, antifungal and Pneumocystis jirovecii pneumonia (PJP) prophylaxis).
4. Intolerance of all trial antibiotic options in either arm A or arm B.
5. Communication, compliance or logistical issues that are likely to limit patient's ability to take prophylactic or emergency antibiotics, or to obtain urgent medical attention for symptoms of infection.
6. Pregnant or breastfeeding.
7. Severe renal impairment (estimated or measured creatinine clearance of less than 30 mL/min).
8. Previous splenectomy.
9. Previous participation in this trial.
10. Treating team deems enrolment in the study is not in the best interests of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS), defined as time from randomisation until occurrence of a Grade 3 or higher infection (as defined by CTCAE Version 5), or death from any cause. | 12 months following randomisation

SECONDARY OUTCOMES:
Proportion of patients who develop at least 1 Grade 3 or higher infection(s) from randomisation to 12 months. | 12 months following randomisation
Proportion of patients with one or more clinically documented infections (symptoms/signs of infection requiring antimicrobial treatment) to 12 months. | 12 months following randomisation
Number of clinically documented infections (symptoms/signs of infection requiring antimicrobial treatment) to 12 months. Data collected from medical records will inform this outcome measure. | 12 months following randomisation
Proportion of patients with one or more microbiologically documented bacterial infections. | 12 months following randomisation
Number of microbiologically documented bacterial infections. | 12 months following randomisation
Time free from hospitalisation and antimicrobials with therapeutic intent. | 12 months following randomisation
Proportion of patients with one or more treatment-related adverse events | 12 months following randomisation
Number of treatment-related adverse events. | 12 months following randomisation
Proportion of patients with fluoroquinolone resistant organisms, co-trimoxazole resistant organisms, extended spectrum beta lactamases or multidrug resistant organisms isolated. | 12 months following randomisation
Number of infections with fluoroquinolone resistant organisms, co-trimoxazole resistant organisms, extended spectrum beta lactamases or multidrug resistant organisms isolated. | 12 months following randomisation
Quality of Life (QoL) measured at randomisation then 3, 6, 9 and 12 months | Randomisation and 3, 6, 9 and 12 months following randomisation.
  QoL will be assessed using the EORTC QLQ-C30 questionnaire.
Quality of Life (QoL) measured at randomisation then 3, 6, 9 and 12 months | Randomisation and 3, 6, 9 and 12 months following randomisation.
  QoL will be assessed using the Functional Assessment of Cancer Therapy - Neutropenia (FACT-N) questionnaire.
Quality of Life (QoL) measured at randomisation then 3, 6, 9 and 12 months | Randomisation and 3, 6, 9 and 12 months following randomisation.
  QoL will be assessed using the EQ-5D-5L questionnaire.
Costs associated with allocated treatment arm and infections during study | 12 months following randomisation
  Costs associated with each treatment arm with be aggregated into Australian dollars. Aggregate costs will be calculated based on the following data sources: medical records, infection-related hospitalisations (using unit costs based on unlinked data from the Victorian Admitted Episodes Dataset, Victorian Emergency Minimum Dataset and the Victorian Cost Data Collection), Medicare Benefits Scheme (MBS), Pharmaceutical Benefits Scheme (PBS) and Australian Immunisation Registry (AIR) data.
Cost effectiveness of the allocated treatment arm | 12 months following randomisation
  Differences in costs and Quality Adjusted Life Years (QALYs) for each of the treatment arms will be aggregated into a cost effectiveness ratio. The following data sources will be used to calculate this outcome measure: the EORTC QLQ-C30 questionnaire will be used to calculate QALYS. Costs will be calculated based on the following data sources: medical records, infection-related hospitalisations (using unit costs based on unlinked data from the Victorian Admitted Episodes Dataset, Victorian Emergency Minimum Dataset and the Victorian Cost Data Collection), Medicare Benefits Scheme (MBS), Pharmaceutical Benefits Scheme (PBS) and Australian Immunisation Registry (AIR) data.
Trough IgG level at 3, 6, 9 and 12 months from baseline. | 3, 6, 9 and 12 months from baseline
Proportion of patients in immunoglobulin cessation treatment arms who restart Ig over 12 months. | 12 months following randomisation
Covid anti-spike protein levels at baseline, 3, 6, 9, and 12 months. | 3, 6, 9 and 12 months following baseline

CONTACTS AND LOCATIONS:
Overall Officials: Prof Erica Wood, Principal Investigator — Monash University; Prof Zoe McQuilten, Principal Investigator — Monash University
Locations (7):
- Australia (7):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Concord Hospital, Concord, New South Wales
  - Royal North Shore, St Leonards, New South Wales
  - Monash Medical Centre, Clayton, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Sunshine Hospital, St Albans, Victoria

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be publicly available. Data will only be presented as a whole, no individual data will be published or presented.